CLINICAL TRIAL: NCT04740983
Title: The Study of Efficacy and Safety of UV Forecasting Based Heliotherapy For Psoriasis in Bangkok, Thailand: A Split-side Pilot Study
Brief Title: Ultraviolet Radiation Forecasting Based Heliotherapy For Psoriasis in Bangkok, Thailand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Einapak Boontaveeyuwat, MD, Consultant dermatologist, Dr., Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 500/62
Record Dates: First submitted 2020-05-23; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis Vulgaris
Keywords: Heliotherapy; sun-bathing; psoriasis; ultraviolet radiation; forecasting; Thailand
MeSH Terms: conditions — Psoriasis | interventions — Heliotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heliotherapy (Experimental): will receive 16-week heliotherapy regimen based on the predicted anti psoriasis effective irradiance values along with olive oil (in-house formulation)
  Interventions: Other: Heliotherapy (a sole sun-bathing)
- Control (No Intervention): only will receive olive oil (in-house formulation)

INTERVENTIONS:
Other: Heliotherapy (a sole sun-bathing) — 16-week heliotherapy regimen based on the predicted anti psoriasis effective irradiance values.
  Arms: Heliotherapy

SUMMARY:
Due to limited number of phototherapy centres and shortage of qualified phototherapy practitioners, heliotherapy has become a promising treatment alternative in Thailand where patients effortlessly receive supervised sun-bathing treatments from their homes whenever they are convenient. We used newly designed deep neural network UV forecasting model developed by using our 10 year-retrospective Solar UV irradiance (280-400 nm) retrieved from a ground based platform at Atmosperic laboratory, Silpakorn University, Nakhon Pathom, Thailand (13.82N 100.04E, 30 m above mean sea level). This model achieved a next-day forecast error of less than 12% which has been the most accurate prediction to date. We designed our 10week heliotherapy regimen based on the predicted anti psoriasis effective irradiance values. We studied efficacy and safety of the 12-week heliotherapy regimen for psoriasis on only ruled acceptable clear sky days in Bangkok, Thailand

DETAILED DESCRIPTION:
We studied efficacy and safety of the 16-week heliotherapy regimen for psoriasis on only ruled acceptable clear sky days in Bangkok, Thailand

ELIGIBILITY:
Inclusion Criteria:

* A psoriasis patient who indicate to have phototherapy and have lesional plagues systemically either on the front-back or left-right.
* A participant is based in Bangkok
* A participant is capable to understand and learn how to use our in-house assembled UV metre and web-based heliotherapy platform.

Exclusion Criteria:

* A participant has any sun-sensitive conditions including photo-aggravated photodermatoses and on photosentisitive drug treatments.
* Breast-feeding, pregnant individuals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Targeted PASI score | 16 weeks
  PASI score for targeted plagues will be evaluated by two independent dermatologists (EB, PA) from standard digital photographs.

SECONDARY OUTCOMES:
Incidence of possible acute side effects after sun bathing | 16 weeks
  Potential acute effects of the exposure of full-spectrum solar radiation